CLINICAL TRIAL: NCT02970916
Title: A Phase II Trial to Assess FOLFIRI+Aflibercept Efficacy in Patients With Oxaliplatin-pretreated Metastatic Colorectal Cancer With or Without ACE Polymorphisms
Brief Title: Phase II Trial to Assess FOLFIRI+Aflibercept Efficacy in Patients With Oxaliplatin-pretreated Metastatic Colorectal Cancer With or Without ACE Polymorphisms
Acronym: POLAF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-16-02
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; FOLFIRI; aflibercept; oxaliplatin; ACE polymorphisms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI+aflibercept (Experimental)
  Interventions: Drug: FOLFIRI+aflibercept

INTERVENTIONS:
Drug: FOLFIRI+aflibercept — Aflibercept: 4 mg/kg administered intravenous infusion on day 1
  FOLFIRI regimen immediately after aflibercept:
  Irinotecan:180 mg/m2 intravenous infusion, folinic acid (dl racemic): 400 mg/m2 intravenous infusion, followed by 5-fluorouracil (5-FU): 400 mg/m2 intravenous bolus, followed by 5-FU: 2400 mg/m2 continuous intravenous infusion over 46 hours.
  * folinic acid: 400 mg/m² (racémic) or 200 mg/m² (L-form)

SUMMARY:
The purpose of this study is to assess FOLFIRI+aflibercept efficacy in patients with or without ACE polymorphisms in terms of Progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically proven adenocarcinoma of the colon and/or rectum,
3. Metastatic disease confirmed.
4. Existence of at least one measurable unidimensional lesion using CT or MRI based on the RECIST criteria, version 1.1
5. Patients with metastatic colorectal cancer (mCRC) that is resistant to or has progressed after an oxaliplatin-containing regimen.
6. Age ≥18 years
7. World Health Organization (WHO) Performance status (PS) 0-2,
8. Hematological status: neutrophils (ANC) ≥1.5x109 /L; platelets ≥100x109 /L; haemoglobin ≥9g/dL
9. Adequate renal function: serum creatinine level < 1.5 x ULN
10. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase (ALP) <5xULN
11. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour.
12. Regular follow-up feasible.
13. For female patients of childbearing potential, negative serum pregnancy test
14. Female patients must commit to using reliable and appropriate methods of contraception until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial.

Exclusion Criteria:

1. Uncontrolled hypercalcemia,
2. Pre-existing permanent neuropathy (NCI grade >2)
3. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive ncephalopathy,
4. Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
5. Treatment with any other investigational medicinal product within 28 days prior to study entry.
6. Other serious and uncontrolled non-malignant disease,
7. History or evidence upon physical examination of CNS metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy),
8. Known Gilbert's syndrome
9. Intolerance to atropine sulfate or loperamide
10. Known dihydropyrimidine dehydrogenase deficiency
11. Treatment with CYP3A4 inducers unless discontinued > 7 days prior to inclusion
12. Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis.
13. Other concomitant or previous malignancy, except: i/ adequately treated insitu carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
14. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
15. Pregnant or breastfeeding women,
16. Patients with known allergy to any excipient to study drugs,
17. History of myocardial infarction and/or stroke within 6 months prior to inclusion, NYHA class III and IV congestive heart failure
18. Bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
FOLFIRI+aflibercept efficacy in terms of Progression-free survival (PFS) with or without ACE polymorphisms. | 30 months

SECONDARY OUTCOMES:
Progression free survival (PFS) with or without AGTR1 polymorphisms, according Serum-level sACE | 30 months
Objective Response Rate (ORR) with or without ACE polymorphisms, AGTR1 polymorphisms, according Serum-level sACE | 30 months
Disease Control Rate (DCR) with or without ACE polymorphisms, AGTR1 polymorphisms, according Serum-level sACE | 30 months
Time to progression (TP) with or without ACE polymorphisms, AGTR1 polymorphisms, according Serum-level sACE | 30 months
Time to treatment failure (TTF) with or without ACE polymorphisms, AGTR1 polymorphisms, according Serum-level sACE | 30 months
Overall survival (OS) with or without ACE polymorphisms, AGTR1 polymorphisms, according Serum-level sACE | 30 months
Number of participants with adverse events as assessed by CTCAE v4.0. | 30 months

OTHER OUTCOMES:
Plasma VEGF levels circulating and their correlation with tumour-efficacy parameters (ORR, PFS and OS) | 30 months
Other biomarkers in serum and tumour tissue associated with cell and tumour growth and/or involved in the mechanism of action of FOLFIRI+aflibercept and their correlation with tumour-efficacy parameters (ORR, PFS and OS) | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Aranda, MD-PhD, Study Chair — Hospital Universitario Reina Sofía; Auxiliadora Gómez, MD-PhD, Study Chair — Hospital Universitario Reina Sofía
Locations (1):
- Spanish Cooperative Group for the Treatment of Digestive Tumors, Madrona, Spain